CLINICAL TRIAL: NCT04164069
Title: A Phase Ib Adaptive Study Dasatinib for the Prevention of Oxaliplatin-Induced Neuropathy in Patients With Metastatic Gastrointestinal Cancer Receiving FOLFOX Chemotherapy With or Without Bevacizumab
Brief Title: Dasatinib for the Prevention of Oxaliplatin-Induced Neuropathy in Patients With Metastatic Gastrointestinal Cancer Receiving FOLFOX Chemotherapy With or Without Bevacizumab
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Anne Noonan (Other)
Responsible Party: Sponsor-Investigator, Anne Noonan, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OSU-19067; NCI-2019-04723 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2019-10-11; First posted 2019-11-15 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-04

CONDITIONS: Advanced Colorectal Carcinoma; Metastatic Colorectal Carcinoma; Stage IV Colorectal Cancer AJCC v8; Stage IVA Colorectal Cancer AJCC v8; Stage IVB Colorectal Cancer AJCC v8; Stage IVC Colorectal Cancer AJCC v8; Stage II Colon Cancer; Stage II Rectal Cancer; Stage III Colon Cancer; Stage III Rectal Cancer; Esophageal Cancer; Pancreatic Cancer; Bile Duct Cancer; Gastric Cancer; Gall Bladder Cancer; Small Bowel Adenocarcinoma
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Esophageal Neoplasms; Pancreatic Neoplasms; Bile Duct Neoplasms; Stomach Neoplasms; Gallbladder Neoplasms | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Dasatinib; Fluorouracil; dehydroftorafur; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Prevention (dasatinib, mFOLFOX, bevacizumab) (Experimental): Patients receive oxaliplatin IV over 2 hours, leucovorin IV over 2 hours, fluorouracil slow IV push over 2-4 minutes followed by continuous infusion over 46 hours on days 1 and 15. Patients also receive dasatinib PO QD on days 14, 15, and 28 of cycle 1 and day 1 of cycle 2. Patients may receive bevacizumab IV over 30 minutes on days 1 and 15. Treatment repeats every 28 days for up to cycle 3 day 1 in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Drug: Dasatinib; Drug: Fluorouracil; Drug: Leucovorin; Drug: Leucovorin Calcium; Drug: Oxaliplatin; Other: Quality-of-Life Assessment

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab awwb; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; BP102; BP102 Biosimilar; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501
Drug: Dasatinib — Given PO
  Other Names: BMS-354825; Dasatinib Hydrate; Dasatinib Monohydrate; Sprycel
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-FU; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Drug: Leucovorin — Given IV
  Other Names: Folinic acid
Drug: Leucovorin Calcium — Given IV
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; citrovorum factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; JM-83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; SR-96669
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase Ib trial studies side effects and best dose of dasatinib in preventing oxaliplatin-induced peripheral neuropathy in patients with gastrointestinal cancers who are receiving FOLFOX regimen with or without bevacizumab. Drugs used in chemotherapy, such as leucovorin, fluorouracil, and oxaliplatin (FOLFOX regimen), work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. However, the buildup of oxaliplatin in the cranial nerves can result in damage or the nerves. Dasatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Blocking these enzymes may reduce oxaliplatin-induced peripheral neuropathy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the recommended phase 2 dose (RP2D) of dasatinib in combination with oxaliplatin and fluorouracil (5FU) (modified version 6 regimen of leucovorin, fluorouracil and oxaliplatin [mFOLFOX6]) with or without bevacizumab in patients with colon, rectal or other GI cancer, defined as the lowest intermittent dose of dasatinib that affects serum biomarkers of OCT2 without influencing the pharmacokinetic properties of oxaliplatin.

II. To determine the toxicity profile (based on Chemotherapy-Induced Peripheral Neuropathy [CIPN]20 and Common Terminology Criteria for Adverse Events [CTCAE] version [v.] 5.0) of dasatinib in combination with oxaliplatin/5-FU/bevacizumab in patients with colorectal cancer or other GI cancer.

SECONDARY OBJECTIVES:

I. To evaluate the influence of dasatinib on the pharmacokinetics of oxaliplatin and vice versa in these patients.

OUTLINE: This is a dose-escalation study of dasatinib.

Patients receive oxaliplatin intravenously (IV) over 2 hours, leucovorin IV over 2 hours, fluorouracil slow IV push over 2-4 minutes followed by continuous infusion over 46 hours on days 1 and 15. Patients also receive dasatinib orally (PO) once daily (QD) on days 14, 15, and 28 of cycle 1 and day 1 of cycle 2. Patients may receive bevacizumab IV over 30 minutes on days 1 and 15. Treatment repeats every 28 days for up to cycle 3 day 1 in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed confirmed stage II, III or IV colon or rectal cancer and other gastrointestinal (GI) cancers (e.g. pancreas, esophagogastric, bile duct, small bowel cancers etc) who are candidates for mFOLFOX6, with or without bevacizumab therapy. Pathological confirmation of colon,rectal or other GI cancer is required. Patients may have had prior therapy for GI cancer.
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* Platelets >= 100 x 10^9/L
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 x upper limit of normal (ULN) unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants
* Activated partial thromboplastin time (aPTT) =< 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Serum creatinine: =< 1.5 x upper limit of normal (ULN), or measured or calculated creatinine clearance (estimated by Cockcroft-Gault formula or measured ) >= 50 mL/min urine protein:creatinine (UPC) < 2
* Total bilirubin =< 2 x ULN
* Aspartate aminotransferase (AST, serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT, serum glutamate pyruvate transaminase [SGPT]) =< 3 x ULN, unless evidence of liver metastases, then AST/alanine aminotransferase (ALT) =< 5 x ULN
* Blood pressure (if receiving bevacizumab): systolic blood pressure (SBP) > 150 or diastolic blood pressure (DBP) > 100
* Serum potassium and magnesium within the institution normal range.
* Corrected QT (QTc) interval =< 450 mSec
* Women of child-bearing potential must agree to use adequate contraception prior to study entry, for the duration of study participation and for 3 months after completion of study treatment administration
* Prior chemotherapy in the adjuvant or metastatic setting is allowed including prior exposure to oxaliplatin in the adjuvant setting for colorectal cancer or other GI cancer as long as neuropathy is grade 1 or less.
* Pre-existing neuropathy is allowed as long as it is grade 1 or less.

Exclusion Criteria:

* Treatment with any other investigational agents within 4 weeks or 5 half-lives (whichever is longer) prior to the first dose of dasatinib
* Gastrointestinal (GI) disease or impairment of GI function that is likely to significantly alter the absorption of dasatinib
* Use of potent OCT2 and/or CYP3A4 inhibitors if treatment cannot be either safely discontinued or switched to a different medication prior to starting dasatinib
* Concurrent cetuximab panitumumab or any other biological/targeted agent.
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, known human immunodeficiency virus (HIV) diagnosis if receiving combination antiretroviral therapy, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations, including psychotic disorders, dementia and substance use disorders, that would limit compliance with study requirements
* Because there is an unknown potential risk for adverse events in nursing infants secondary to treatment of the mother with dasatinib and/or oxaliplatin, breastfeeding should be discontinued
* Inability to understand and sign informed consent
* Any other condition that in the opinion of the investigators would make the study therapy unsafe

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
Recommended phase II dose (RP2D) of dasatinib | Up to 14 days
  The RP2D will be defined as the lowest intermittent dose of dasatinib that affects serum biomarkers of OCT2 without influencing the pharmacokinetic properties of oxaliplatin.
Incidence of adverse events | At the end of Cycle 1 (cycle length is 28 days)
  The dose-limiting toxicity and toxicity profile will be based using the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 and Chemotherapy-Induced Peripheral Neuropathy (CIPN) 20. Toxicity will be defined as adverse events deemed to be at least possibly related to dasatinib treatment. Adverse events and toxicities will be summarized by dose level, and will tabulate these events by type and severity. Will summarize the numbers of patients who required dose reductions in dasatinib or oxaliplatin and the cumulative doses received. The CIPN20 will be measured in these subjects, and will be summarized within and across dose levels, and will be used to support and inform assumptions for a subsequent phase 2 trial.

OTHER OUTCOMES:
Dasatinib on pharmacokinetics (PK) of oxaliplatin | Baseline, days 1, 2, and 14
  Objective is to evaluate the influence of dasatinib on the pharmacokinetics of oxaliplatin and vice versa. Oxaliplatin PK will be measured at pre-dose, 1 hour, immediately prior to end of infusion of oxaliplatin, and 0.5, 1, 2, 4 hours after end of infusion on day 1; Dasatinib PK will be measured at pre-dose and 0.5, 1.5, 2.5, 3, 4.5, and 6.5 hours after taking dasatinib on day 14; PK of dasatinib and oxaliplatin will be measured on day 15 pre-dose of dasatinib, prior to starting oxaliplatin infusion, 1 hour after start of oxaliplatin infusion, immediately prior to end of infusion with oxaliplatin, and at 0.5, 1, 2, 4 hours after end of oxaliplatin infusion. PK parameters calculated using standard non-compartmental methods, and non-linear mixed effect models will be created to inform the use of limited-sampling strategies for subsequent confirmatory studies. Area Under the Curve [AUC] will be calculated for each drug Oxaliplatin - ug x h/ml and Dasatinib- ng x h/ml

CONTACTS AND LOCATIONS:
Overall Officials: Anne M Noonan, MBBChBAO, MSc, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stage TB, Hu S, Sparreboom A, Kroetz DL. Role for Drug Transporters in Chemotherapy-Induced Peripheral Neuropathy. Clin Transl Sci. 2021 Mar;14(2):460-467. doi: 10.1111/cts.12915. Epub 2020 Nov 9. PMID 33142018
- See also: The Jamesline — http://cancer.osu.edu

DOCUMENTS (1):
  • Informed Consent Form (2021-10-28): https://cdn.clinicaltrials.gov/large-docs/69/NCT04164069/ICF_000.pdf